CLINICAL TRIAL: NCT02653846
Title: Correlation of Liver and Spleen Stifness as Assesed by Real Time 2-Dimensional Shear Wave Elastography With Severity of Portal Hypertension and Clinical Outcomes in Patients With Compensated Advanced Chronic Liver Disease
Brief Title: Correlation of Liver and Spleen Stiffness by RT-2D-SWE and Severity of Portal Hypertension by HVPG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Ivica Grgurevic, MD, Assist. prof. Ivica Grgurevic, MD, PhD, FEBGH, University Hospital Dubrava
Other Study IDs: KBD-IG-LS/SSvsHVPG
Record Dates: First submitted 2015-12-31; First posted 2016-01-12 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: RT-2D-SWE measurement — measurement of liver and spleen stiffness by ultrasound real-time 2D shear wave elastography (SWE™)
Procedure: HVPG measurement — assessment of portal hypertension assessed by hepatic venous pressure gradient measurement

SUMMARY:
Portal hypertension (PH) results from the increase of portal flow resistance in fibrotic tissue of the liver in patients with chronic liver diseases, leading to complications such as varices formation and variceal bleeding, ascites formation, spleenomegaly and hypersplenismus, systemic haemodynamic disorders and porto-systemic shunts formation. Early detection of PH in patients with chronic liver diseases is clinically important as it should change patient management in order to prevent the formation/onset or recurrence of PH complications. Hepatic venous pressure gradient (HVPG) measurement is the gold standard for the assessment of the severity of PH. However, it is an invasive method with its risks, and relatively costly. On the other hand transient elastography (TE) emerged as a non-invasive, easy, safe and low cost method with the potential to assess the severity of PH, as liver stiffness (LS) and spleen stiffens (SS) measured by TE showed very good correlation with HVPG. Real-time 2D shear wave elastography (RT-2D-SWE) is an ultrasound elastography method reliable for non-invasive assessment of fibrosis stage especially in chronic viral hepatitis, but only preliminary data exist on the correlation of RT-2D-SWE measured LS/SS with and HVPG. In this study we hypothesized that LS and SS measured by RT-2D-SWE correlate with HVPG enabling RT-2D-SWE to be used for the assessment of severity of PH. The primary aim of this study is to analyse correlation between LS and SS as assessed by RT-2D-SWE and TE with the grade of portal hypertension as assessed by HVPG. The secondary aims are: 1) to analyse clinical outcomes of these patients in order to determine if LS and/or SS as assessed by RT-2D-SWE might predict adverse outcomes (liver decompensation, death or HCC development), and 2) to compare clinical performance (AUC) of RT-2D-SWE and TE for the assessment of the PH severity as well as for predicting clinical outcomes. Patients with suspicion of having compensated advanced chronic liver disease (cACLD) as assesed by non-invasive methods (transabdominal ultrasound, laboratory findings, FIB-4 and APRI score, and LS measurements by TE), will be included. Since positive predictive value of non-invasive methods for cirrhosis is generally not very reliable, these patients will be offered transjugular liver biopsy and HVPG measurements as gold-standard methods to define the stage of liver disease and severity of PH. These patients will undergo LS and SS measurements by RT-2D-SWE on Aixplorer SuperSonic Imagine ultrasound system and HVPG measurements as well, with transjugular liver biopsy performed during the same session. After SWE™ and HVPG measurement, 5-year follow-up is planned, including standard surveillance: laboratory findings, transabdominal US every six months and upper-GI endoscopy according to relevant guidelines, as well as treatment according to relevant guidelines as indicated: beta blockers, endoscopic variceal ligation, etiologic treatment and dietary measures. Appropriate statistical analysis will be undertaken after the enrollment period, as well as after follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspicion of having cACLD as assessed by transabdominal ultrasound, laboratory findings, FIB-4 and/or APRI score, and/or LS measurements
* patients with chronic liver disease in whom any extrahepatic surgical procedure is planned and in whom it was not possible to exclude cACLD and/or portal hypertension based on non-invasive procedures only
* patients with HCC or other liver tumors on the ground of presumed liver cirrhosis who are under consideration for surgical resection, in whom HVPG is performed in order to reliably exclude clinically significant portal hypertension
* compliance to the study protocol
* signed approval for the diagnostic ultrasound with SWE™ and for transjugular liver biopsy and HVPG measurement

Exclusion Criteria:

* elevated alanine aminotransferase (ALT) values > 5 x upper limit of normal (ULN)
* obstructive jaundice
* congestive heart failure
* sepsis
* thrombosis of right jugular vein
* thrombosis of hepatic veins
* hydatid cyst
* cholangitis
* absence of cooperation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients and inpatients in a tertiary care hospital 1) with suspicion of having compensated advanced chronic liver disease (cACLD) as assessed by transabdominal ultrasound, laboratory findings, FIB-4 and/or APRI score, and/or LS measurements by TE; 2) patients with chronic liver disease in whom any extrahepatic surgical procedure is planned and in whom it was not possible to exclude cACLD and/or portal hypertension based on non-invasive procedures only; 3) patients with HCC or other liver tumors on the ground of presumed liver cirrhosis who are under consideration for surgical resection, in whom HVPG is performed in order to reliably exclude clinically significant portal hypertension
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
liver and spleen stiffness | at the time of enrollment
  liver and spleen stiffness expressed in kPa, measured by real-time 2D shear wave elastography (SWE™) on Aixplorer® ultrasound machine from SuperSonic Imagine, Aix-en-Provence, France
HVPG | within one week of enrollment
  severity of portal hypertension assessed by hepatic venous pressure gradient (HVPG) measurements

SECONDARY OUTCOMES:
development of hepatic decompensation | during follow-up period of 5 years
  hepatic decompensation defined as: onset of icterus, onset of ascites diagnosed by transabdominal ultrasonud or CT scan, onset of portal encephalophaty diagnosed clinically, episode of variceal bleeding confirmed endoscopically
Hepatocellular carcinoma (HCC) development | during follow-up period of 5 years
  conformed by contrast MDCT and/or MRI and/or tumor biopsy
mortality | during follow-up period of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ivica Grgurevic, MD, PhD, Principal Investigator — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berzigotti A, Seijo S, Arena U, Abraldes JG, Vizzutti F, Garcia-Pagan JC, Pinzani M, Bosch J. Elastography, spleen size, and platelet count identify portal hypertension in patients with compensated cirrhosis. Gastroenterology. 2013 Jan;144(1):102-111.e1. doi: 10.1053/j.gastro.2012.10.001. Epub 2012 Oct 8. PMID 23058320
- [Background] Augustin S, Millan L, Gonzalez A, Martell M, Gelabert A, Segarra A, Serres X, Esteban R, Genesca J. Detection of early portal hypertension with routine data and liver stiffness in patients with asymptomatic liver disease: a prospective study. J Hepatol. 2014 Mar;60(3):561-9. doi: 10.1016/j.jhep.2013.10.027. Epub 2013 Nov 6. PMID 24211744
- [Background] Vergniol J, Foucher J, Terrebonne E, Bernard PH, le Bail B, Merrouche W, Couzigou P, de Ledinghen V. Noninvasive tests for fibrosis and liver stiffness predict 5-year outcomes of patients with chronic hepatitis C. Gastroenterology. 2011 Jun;140(7):1970-9, 1979.e1-3. doi: 10.1053/j.gastro.2011.02.058. Epub 2011 Mar 2. PMID 21376047
- [Background] Colecchia A, Montrone L, Scaioli E, Bacchi-Reggiani ML, Colli A, Casazza G, Schiumerini R, Turco L, Di Biase AR, Mazzella G, Marzi L, Arena U, Pinzani M, Festi D. Measurement of spleen stiffness to evaluate portal hypertension and the presence of esophageal varices in patients with HCV-related cirrhosis. Gastroenterology. 2012 Sep;143(3):646-654. doi: 10.1053/j.gastro.2012.05.035. Epub 2012 May 27. PMID 22643348
- [Background] Colecchia A, Colli A, Casazza G, Mandolesi D, Schiumerini R, Reggiani LB, Marasco G, Taddia M, Lisotti A, Mazzella G, Di Biase AR, Golfieri R, Pinzani M, Festi D. Spleen stiffness measurement can predict clinical complications in compensated HCV-related cirrhosis: a prospective study. J Hepatol. 2014 Jun;60(6):1158-64. doi: 10.1016/j.jhep.2014.02.024. Epub 2014 Mar 6. PMID 24607624
- [Background] Behrens G, Ferral H. Transjugular liver biopsy. Semin Intervent Radiol. 2012 Jun;29(2):111-7. doi: 10.1055/s-0032-1312572. PMID 23729981
- [Background] Dohan A, Guerrache Y, Boudiaf M, Gavini JP, Kaci R, Soyer P. Transjugular liver biopsy: indications, technique and results. Diagn Interv Imaging. 2014 Jan;95(1):11-5. doi: 10.1016/j.diii.2013.08.009. Epub 2013 Sep 3. PMID 24007769